CLINICAL TRIAL: NCT04574934
Title: Effect of Aquatic Therapy on Pulmonary Functions in Patients With Muscular Dystrophy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammed E. Ali, Ph. D Candidate., Principal Investigator, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002574
Record Dates: First submitted 2020-08-05; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Muscular Dystrophy
Keywords: Aquatic Therapy; pulmonary Functions; muscular dystrophy
MeSH Terms: conditions — Muscular Dystrophies | interventions — Aquatic Therapy

STUDY DESIGN:
Intervention Model Description: Thirty patients with muscular dystrophy were enrolled in this study and were assessed for eligibility. Their age ranged from four and forty years. They were assigned randomly into two equal groups. Group (A) study group received the traditional physical therapy program plus aquatic therapy. And the group (B) control group received traditional physical therapy program only. All patients will receive sessions two times/week for three successive months. Pulmonary function test was used to assess pulmonary functions pre and post-intervention. All patients were assisted before and after three months of intervention.
Who Masked: Outcomes Assessor
Masking Description: Blinding process to participants and care providers was impossible because of intervention therapy. We analyzed data by an impartial statistician (outcomes assessor), referring to each arm with an encoded name: Group A (study group) and Group B (control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the study group (Experimental): study group received the traditional physical therapy program plus aquatic therapy
  Interventions: Other: aquatic therapy
- the control group (No Intervention): control group received traditional physical therapy program only.

INTERVENTIONS:
Other: aquatic therapy — Aquatic therapy refers to water-based treatments or exercises of therapeutic intent, in particular for relaxation, fitness, and physical rehabilitation. Treatments and exercises are performed while floating, partially submerged, or fully submerged in water. Many aquatic therapy procedures require constant attendance by a trained therapist and are performed in a specialized temperature-controlled pool. Rehabilitation commonly focuses on improving the physical function associated with illness, injury, or disability
  Arms: the study group

SUMMARY:
This study aimed to assess the efficacy of aquatic therapy on pulmonary functions in patients with muscular dystrophy.

DETAILED DESCRIPTION:
Muscular dystrophy (MD) is a group of muscle diseases that results in increasing weakening and breakdown of skeletal muscles over time. The disorders differ in which muscles are primarily affected, the degree of weakness, how fast they worsen, and when symptoms begin. Many people will eventually become unable to walk. Some types are also associated with problems in other organs. The muscular dystrophy group contains thirty different genetic disorders that are usually classified into nine main categories or types.

The signs and symptoms consistent with muscular dystrophy are: progressive muscular wasting, poor balance, scoliosis (curvature of the spine and the back), progressive inability to walk, waddling gait, Calf deformation, Limited range of movement,respiratory difficulty, cardiomyopathy and muscle spasms

ELIGIBILITY:
Inclusion Criteria:

* Their age will ranging from four to forty years.
* Patients participated in this study will from both sexes.
* All patients will able to walk supported or unsupported by the therapist.
* All patients will able to follow the instructions during testing and training.
* All patients had no fixed contractures or deformities at the lower limb.

Exclusion Criteria:

* Patients with visual or auditory problems.
* Patients with structural joints deformities of the lower limbs.
* Patients with convulsions and fixed contractures.
* Uncooperative Patient.

Ages: 4 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | Forced Vital Capacity (FVC) will be assessed at day 0.
  Forced vital capacity (FVC) is the amount of air that can be forcibly exhaled from your lungs after taking the deepest breath possible, as measured by spirometry.
Forced Vital Capacity (FVC) | Forced Vital Capacity (FVC) will be assessed at day 90.
  Forced vital capacity (FVC) is the amount of air that can be forcibly exhaled from your lungs after taking the deepest breath possible, as measured by spirometry.
Forced Expiratory Volume (FEV1) | Forced Expiratory Volume (FEV1) will be assessed at day 0.
  Forced expiratory volume in one second (FEV1) is a measurement of your ability to expel air from your lungs. More specifically, and as its name suggests, it is the amount that is exhaled in the first second of purposefully trying to breathe out as much air as possible.
Forced Expiratory Volume (FEV1) | Forced Expiratory Volume (FEV1) will be assessed at day 90.
  Forced expiratory volume in one second (FEV1) is a measurement of your ability to expel air from your lungs. More specifically, and as its name suggests, it is the amount that is exhaled in the first second of purposefully trying to breathe out as much air as possible.
Forced Expiratory Volume/Forced Vital Capacity Ratio (FEV1/FVC ratio) | Forced Expiratory Volume/Forced Vital Capacity Ratio (FEV1/FVC ratio) will be assessed at day 0.
  is a calculated ratio used in the diagnosis of obstructive and restrictive lung disease.[2][3] It represents the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration (FEV1) to the full, forced vital capacity (FVC).[4] The result of this ratio is expressed as FEV1%. Normal values are approximately 75%.[5] Predicted normal values can be calculated online and depend on age, sex, height, and ethnicity as well as the research study that they are based upon. A derived value of FEV1% is FEV1% predicted, which is defined as FEV1% of the patient divided by the average FEV1% in the population for any person of similar age, sex, and body composition.
Forced Expiratory Volume/Forced Vital Capacity Ratio (FEV1/FVC ratio) | Forced Expiratory Volume/Forced Vital Capacity Ratio (FEV1/FVC ratio) will be assessed at day 90.
  is a calculated ratio used in the diagnosis of obstructive and restrictive lung disease.[2][3] It represents the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration (FEV1) to the full, forced vital capacity (FVC).[4] The result of this ratio is expressed as FEV1%. Normal values are approximately 75%.[5] Predicted normal values can be calculated online and depend on age, sex, height, and ethnicity as well as the research study that they are based upon. A derived value of FEV1% is FEV1% predicted, which is defined as FEV1% of the patient divided by the average FEV1% in the population for any person of similar age, sex, and body composition.

CONTACTS AND LOCATIONS:
Overall Officials: Nehad A. Abo-zaid, Ph.D, Principal Investigator — South Valley University; Mohammed E. Ali, Ph.D student, Principal Investigator — South Valley University
Locations (1):
- South Valley University, Faculty of Physical Therapy, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eagle M. Report on the muscular dystrophy campaign workshop: exercise in neuromuscular diseases Newcastle, January 2002. Neuromuscul Disord. 2002 Dec;12(10):975-83. doi: 10.1016/s0960-8966(02)00136-0. No abstract available. PMID 12467755
- [Background] Bach JR, Martinez D. Duchenne muscular dystrophy: continuous noninvasive ventilatory support prolongs survival. Respir Care. 2011 Jun;56(6):744-50. doi: 10.4187/respcare.00831. Epub 2011 Feb 11. PMID 21333078
- [Result] Khirani S, Ramirez A, Aubertin G, Boule M, Chemouny C, Forin V, Fauroux B. Respiratory muscle decline in Duchenne muscular dystrophy. Pediatr Pulmonol. 2014 May;49(5):473-81. doi: 10.1002/ppul.22847. Epub 2013 Jul 8. PMID 23836708
- [Result] Fowler WM Jr. Role of physical activity and exercise training in neuromuscular diseases. Am J Phys Med Rehabil. 2002 Nov;81(11 Suppl):S187-95. doi: 10.1097/01.PHM.0000029726.80774.83. PMID 12409823
- [Result] Abresch RT, Carter GT, Han JJ, McDonald CM. Exercise in neuromuscular diseases. Phys Med Rehabil Clin N Am. 2012 Aug;23(3):653-73. doi: 10.1016/j.pmr.2012.06.001. PMID 22938880

DOCUMENTS (1):
  • Study Protocol (2020-09-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT04574934/Prot_000.pdf